CLINICAL TRIAL: NCT04219098
Title: Pain After Preoperative UltraSound Guided Hip Injections for Total Hip Arthroplasty (PUSH)
Acronym: PUSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anne Arundel Health System Research Institute (Other)
Responsible Party: Principal Investigator, Paul King, Director of the Center for Joint Replacement, Anne Arundel Health System Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Designer [1544619
Record Dates: First submitted 2019-12-30; First posted 2020-01-06 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Total Hip Replacement; Arthroplasty
Keywords: THA; THR
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This study is designed to be prospective randomized (1:1) controlled independent trial.
Who Masked: Care Provider, Investigator
Masking Description: Only the surgeon and PA will be aware of the randomization assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Butterfly IQ utilized to inject 10cc prior to surgery the remainder after incision
  Interventions: Procedure: Butterfly IQ
- Control (Active Comparator): Entire injection will be given after initial incision is made.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Procedure: Butterfly IQ — 10ml of solution with .5cc (or one drop) sterile methylene blue will be injected intra-articularly under ultrasound guidance after a sterile prep. The remaining 20ml will be injected into the periarticular tissues after prosthesis implantation before closure.
  Arms: Treatment
Other: Standard of Care — The entire volume will be injected into the periarticular tissues after prosthesis implantation before closure.
  Arms: Control

SUMMARY:
The purpose of the study is to assess the accuracy of Butterfly IQ ultrasound for intra-articular hip injections, and to see if an injection given intra-articular before incision provides any benefit in preemptive pain relief or blood loss reduction.

DETAILED DESCRIPTION:
This study is designed to be prospective randomized (1:1) controlled independent trial. Subjects are male and female, aged 18 and above, who are suitable candidates for either a unilateral (i.e. single) total hip replacement. Subjects that are scheduled with a single, extensively trained Physician Assistant assisting in their surgery will be exclusively included. This is single site study with projected enrollment of 150 subjects

ELIGIBILITY:
Inclusion Criteria

Subjects meeting all of the following specific criteria will be considered for participation in the study:

1. Subject is between 18-80 years of age.
2. Subject is a suitable candidate for total hip replacement.
3. Subject scheduled for surgery with the Butterfly IQ trained PA providing surgical assistance
4. Subject has given voluntary, written informed consent to participate in this clinical investigation and has authorized the transfer of his/her information to AAHS RI
5. Subject, in the opinion of the Clinical Investigator, is able to understand this clinical investigation and is willing and able to perform all study procedure and follow-up visits and co-operate with investigational procedures.
6. Subject must be comfortable with speaking, reading, and understanding questions in English and providing an appropriate response.

Exclusion Criteria

Subjects will be excluded from participation in the study if they meet any of the following criteria:

1. Subject is a woman who is pregnant or lactating
2. Subject from the vulnerable groups: prisoners, adults unable to consent, children, non-English speaking, illiterate, and/or visually impaired)
3. Subject who is not comfortable with speaking, reading, and understanding questions in English and providing an appropriate response.
4. Subject who cannot or refuses to give voluntary, written informed consent to participate in this clinical trial
5. Subject has contraindications for any of the following: Ropivicaine, Epinephrine or Methylene Blue
6. Previous hip surgery
7. History of infection in hip
8. Morbid obesity defined as BMI>40

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Accuracy | Surgery
  Primary objective is to determine the accuracy of the Butterfly IQ portable app based ultrasound device used in intra-articular hip injections determined by patient reported pain ratings using the Patient Reported Outcome Measure Information System (PROMIS) pain rating 0(no pain)- 5 (most pain)

SECONDARY OUTCOMES:
Blood Loss | Postoperative day 1
  Evaluate blood loss as determined by relative change in HCT preoperatively and on the first post-operative day.

CONTACTS AND LOCATIONS:
Locations (1):
- Anne Arundel Medical Center, Annapolis, Maryland, United States

IPD SHARING:
Plan to Share IPD: No